CLINICAL TRIAL: NCT06671080
Title: Upper Extremity Performance, Balance and Core Endurance in Adolescent Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep HOŞBAY, Assistant Professor, Biruni University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: adolescent soccer players
Record Dates: First submitted 2024-10-16; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Sports Physical Therapy
Keywords: Upper Extremity Performance; Balance; Core Endurance; Soccer

STUDY DESIGN:
Intervention Model Description: In the study, quantitative evaluation tests will be conducted and numerical data will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment Group (Experimental): All of the tests planned to be used in the study will be applied to adolescent amateur soccer players who meet the inclusion criteria.
  Interventions: Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test

INTERVENTIONS:
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test — All of these tests planned to be used in the study will be applied to adolescent amateur soccer players who meet the inclusion criteria.
  Other Names: Upper Quarter Y Balance Test; Star Excursion Balance Test; Mcgill Core Endurance Test

SUMMARY:
Soccer is one of the most popular sports in the world with a large number of players under the age of 18. High physical demands, frequent changes in exercise intensity and a large number of movement profiles require optimal physical capacity for both adult and child players in soccer.

Physical Performance Tests (PPT) are used to provide a detailed overview of functional status, to predict injury or to decide on return to sport. Physical performance is assessed using closed or open kinetic chain tests; however, in athletic populations, closed kinetic chain PTs may allow for more comprehensive assessments than open kinetic chain PTs.

The continuity of the kinetic chain is required for biomechanically and kinesiologically correct performance of upper extremity functions during daily life activities. The kinetic chain is a system that enables different body parts to produce and transfer power in coordination. The system creates minimal stress, maximal power generation and transfer in the kinetic chain, thus supporting the movement in the distal segments. In order to ensure minimal loss in power transfer between the extremities and trunk, trunk stabilization with a strong core is required.

Athletic performance can be assessed by functional, agility, speed and power tests involving the extremities or the whole body. According to the kinetic chain theory, a "break in the chain" can lead to a decrease in optimal force production and a decrease in performance. The relationship between balance, strength and endurance parameters can provide a basis for the assessment of injury risks and the development of preventive programs. In the literature, it has been suggested that factors related to strength and functionality of the upper extremity may be related to endurance and performance. The aim of this study was to investigate the relationship between upper extremity performance, balance and core endurance in adolescent soccer players.

DETAILED DESCRIPTION:
Soccer is one of the most popular sports in the world with a large number of players under the age of 18. High physical demands, frequent changes in exercise intensity and a large number of movement profiles require optimal physical capacity for both adult and child players in soccer.

Physical Performance Tests (PPT) are used to provide a detailed overview of functional status, to predict injury or to decide on return to sport. Physical performance is assessed using closed or open kinetic chain tests; however, in athletic populations, closed kinetic chain PTs may allow for more comprehensive assessments than open kinetic chain PTs.

Balance is one of the important factors determining sportive performance. It provides neuromuscular control by integrating central nervous system stimuli from the environment to maintain postural control on unstable surfaces during sports activities. Soccer is often played on unstable surfaces (e.g., jumping on grass, kicking the ball while being blocked by an opponent), and the factors affecting players' balance are greater than in other sports. This suggests that soccer players need to have a more dynamic balance compared to other athletes.

The core is the power center of the body with the abdominal muscles on the front, paraspinal and gluteal muscles on the back, diaphragm on the roof, oblique abdominal muscles on the sides, and pelvic ring on the floor. The core acts as a muscular corset to stabilize the trunk with or without limb movement. Core stability enhances effective control of the trunk and stabilization of posture and provides a fundamental basis for force generation and transmission between the upper and lower extremities.

The continuity of the kinetic chain is required for biomechanically and kinesiologically correct performance of upper extremity functions during daily life activities. The kinetic chain is a system that enables different body parts to produce and transfer power in coordination. The system creates minimal stress, maximal power generation and transfer in the kinetic chain, thus supporting the movement in the distal segments. In order to ensure minimal loss in power transfer between the extremities and trunk, trunk stabilization with a strong core is required.

Athletic performance can be assessed by functional, agility, speed and power tests involving the extremities or the whole body. According to the kinetic chain theory, a "break in the chain" can lead to a decrease in optimal force production and a decrease in performance [16]. The relationship between balance, strength and endurance parameters can provide a basis for the assessment of injury risks and the development of preventive programs. In the literature, it has been suggested that factors related to strength and functionality of the upper extremity may be related to endurance and performance. The aim of this study was to investigate the relationship between upper extremity performance, balance and core endurance in adolescent soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Athletes between the ages of 13-16
* Be actively playing amateur football for at least 1 year in any football team
* Playing soccer regularly for 60 minutes at least 3 days a week

Exclusion Criteria:

* A shoulder problem in the last three months,
* He plays in the goalkeeper position,
* Not having any disease (cardiac, orthopedic or neurological) that may prevent participation in the study,
* Having circulatory problems such as varicose veins,
* Surgical history in the last 6 months,
* Receiving any other physiotherapy treatment,
* The presence of symptoms such as vertigo,
* Presence of complaints in the musculoskeletal system of the elbow, wrist, hand and trunk and lower extremities

Ages: 13 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Amateur male soccer players between the ages of 13-16
Enrollment: 52 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Closed Kinetic Chain Upper Extremity Stability Test | through study completion, an average of 6 months.
  It is used to assess upper extremity strength, endurance and closed kinetic chain. The test is performed as follows: In the push-up position, the distance between the two hands is adjusted to 90 cm, then one hand is extended towards the other hand and the number of repetitions completed within 15 s is recorded. The test is repeated 3 times. A rest period of 45 s is allowed between tests to avoid fatigue caused by high intensity activity (1:3 activity/rest ratio).

SECONDARY OUTCOMES:
Upper Quarter Y Balance Test | through study completion, an average of 6 months.
  The assessment is started in the push-up position with both arms shoulder-width apart. Starting with the non-dominant hand, the maximum distance reached in the medial, inferolateral and superiolateral directions is recorded. To determine upper extremity length, the distance between C7 and the 3rd fingertip is measured in cm in the anatomical position with the shoulder joint in 90° abduction. In cases where the feet are off the ground during the tests, significant flexion of the hip occurs, load is transferred to the reaching arm and the elbow of the stable arm is flexed, the test is considered invalid and the test is restarted.
Star Excursion Balance Test | through study completion, an average of 6 months.
  For the test setup, 4 1.5-meter tape measures are attached to the floor at a 45-degree angle. The athlete is asked to stand on one foot at the intersection point and extend the toe of the other foot in 8 directions (anterior, anterolateral, lateral, posterolateral, posterior, posteromedial, medial and anteromedial). Meanwhile, the person should not lose his/her balance and should not lift the heel of the foot on which he/she is standing off the ground.
Mcgill Core Endurance Test | through study completion, an average of 6 months.
  McGill's trunk muscle endurance tests are used to assess core stability. Trunk flexor endurance test (TFET), trunk extensor endurance test (TEET), bilateral side bridge endurance tests (SBET).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep HOŞBAY, PHD, Study Director — Biruni University
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)